CLINICAL TRIAL: NCT05830383
Title: Application of PDCA Circular Management to Improve Critical Thinking Skills of ICU Nurses Within Five Years of Employment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SYSKY-2023-256-01
Record Dates: First submitted 2023-04-03; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-03

CONDITIONS: PDCA Circular Management
Keywords: PDCA circular management;critical thinking skills

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PDCA circular management (Experimental): The countermeasure 1-ABC rescue training:Clarify the positions and perform their duties; Countermeasure 2-Advanced Life Support (ACLS) training: Clear division of labor and strengthen the cooperation Tune; Countermeasure 3-Objective Structural Clinical Test (OSCE Exam): Objective, orderly, and organized assessment
  Interventions: Behavioral: PDCA circular management

INTERVENTIONS:
Behavioral: PDCA circular management — PDCA circular management means "Plan""Do""Check""Action" four steps

SUMMARY:
Choose about 100 low -age nurses who have been in the ICU in 2022, and conduct a scoring score of the survey and critical thinking skills through the schedule. Based on the survey and scoring results ,Formulate the PDCA circular management process and conduct a judgment of critical thinking skills after intervention.To compare the critical thinking skills survey score before and after.

DETAILED DESCRIPTION:
Through the countermeasure 1-ABC rescue training: Clarify the positions and perform their duties; Countermeasure 2-Advanced Life Support (ACLS) training: Clear division of labor and strengthen the cooperation Tune; Countermeasure 3-Objective Structural Clinical Test (OSCE Exam): Objective, orderly, and organized assessment. The framework and group competitions are evaluated to promote teaching and other measures.The comparison experimental objects use the data of the two questionnaires before and after the PDCA cycle management. Explore the application effect of PDCA circular management within five years of employment.

ELIGIBILITY:
Inclusion Criteria: (1) ICU nurse within five years of joining the ICU

(2) Voluntary participation in this study.

-

Exclusion Criteria:(1) Clinical nurses who have worked for more than 5 years

(2) Involuntary participation in this study.

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-03-27 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
critical thinking | 1 year
  The score of critical thinking skills after interventions

CONTACTS AND LOCATIONS:
Overall Officials: huiying Fuhuiying, Principal Investigator — colleague
Locations (1):
- One Case of Individualized Nursing Plan for Sepsis, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boso CM, van der Merwe AS, Gross J. Critical thinking disposition of nursing students: A quantitative investigation. Nurse Educ Pract. 2021 Aug;55:103167. doi: 10.1016/j.nepr.2021.103167. Epub 2021 Jul 30. PMID 34358855
- [Result] Christodoulakis A, Zografakis Sfakianakis M, Tsiligianni I. Suggestions for overcoming the barriers to critical thinking in nursing. Jpn J Nurs Sci. 2023 Jul;20(3):e12525. doi: 10.1111/jjns.12525. Epub 2023 Feb 8. PMID 36755474